CLINICAL TRIAL: NCT05285410
Title: Observational Study of Telehealth for Remote Endpoint Assessment (OUTREACH)
Brief Title: Observational Study Comparing Home to Office Spirometry
Acronym: OUTREACH
Status: Completed | Type: Observational
Sponsor: Chris Goss (Other)
Collaborators: University of Washington (Other); University of Arkansas (Other); Harvard University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Professor of Medicine and Pediatrics, University of Washington, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: OUTREACH-OB-22
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cystic Fibrosis
Keywords: Telehealth; Spirometry; Cystic Fibrosis; CF; Telemedicine; ZEPHYRx
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal multicenter observational study comparing home to office spirometry and home to office weight and height measurements. The aim of the study is to estimate the accuracy and variability of home spirometric measurements over time, and to assess the feasibility and acceptability of home measurements.

DETAILED DESCRIPTION:
After successful completion of the run-in period, participants will have 3 in-person visits, at which office spirometry will be performed and weight and height measured. Participants will perform home spirometry weekly during the study period. They will also electronically complete a weekly electronic patient reported outcome (ePRO) Within one week of each in-person visit, they will measure height and weight at home and perform home spirometry with virtual coaching by site research staff. They will complete a brief ePRO every 4 weeks regarding acceptability and feasibility of home spirometry in research. Within two weeks after study completion, a purposive subsample will complete an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of a CF diagnosis
* Clinically stable
* ≥6 years of age at Screening Visit
* During the run-in period, performed acceptable home spirometry at least twice without virtually coaching and once with virtually coaching

Exclusion Criteria:

* History of lung transplantation
* Initiation of a highly effective modulator therapy within 2 months before Screening Visit

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited at Cystic Fibrosis Foundation's Therapeutics Development Network study sites
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Difference (bias) in home spirometry compared to office spirometry for 12-week forced expiratory volume in 1 second (FEV1) (% predicted) change | Week 0 to Week 12
  Difference between home and office spirometry estimates of FEV1 (% predicted) change from Week 0 to Week 12 (home estimate - office estimate)
Analytic efficiency of home versus office spirometry for 12-week FEV1 (% predicted) change | Week 0 to Week 12
  Factor by which trial sample size must increase/decrease to maintain a given power going from office to home spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rosenfeld, MD, MPH, Principal Investigator — University of Washington, Seattle Children's Research Institute; Ariel Berlinski, MD, Principal Investigator — University of Arkansas for Med. Sciences, Arkansas Children's Hospital; Andrea Hartzler, PhD, Principal Investigator — University of Washington; Greg Sawicki, MD, MPH, Principal Investigator — Harvard University and Boston Children's Hospital
Locations (19):
- United States (19):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Lenox Hill Hospital Cystic Fibrosis Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - The Adult Cystic Fibrosis Center of Central Texas, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Clinic - Pediatrics, Spokane, Washington
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin